CLINICAL TRIAL: NCT02774642
Title: The Impact of Integrated CBT-I and PE on Sleep and PTSD Outcomes
Brief Title: Integrated CBT-I and PE on Sleep and PTSD Outcomes (Impact Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2120-W; 1lK2Rx002120-01 (Other Grant/Funding Number: Federal Identifier)
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Posttraumatic Stress Disorders; Chronic Insomnia
Keywords: PTSD; insomnia; CBT-I; Prolonged Exposure; Veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTI-PE (Experimental): Integrates the core components of CBT-I and PE in 14 90-minute weekly sessions.
  Interventions: Behavioral: CBTI-PE
- Hygiene-PE (Active Comparator): Uses non-active sleep hygiene to account for the dose response of experimental condition before starting PE. Uses 14 90-minute weekly sessions.
  Interventions: Behavioral: Hygiene-PE

INTERVENTIONS:
Behavioral: CBTI-PE — Integrates CBT-I and PE with the goal of enhancing both insomnia and PTSD outcomes. Integrated treatment will be delivered in 14 90-minute weekly sessions. CBTI-PE starts with VA rollout CBT-I for the first 3 weeks with a focus on the effects of PTSD on insomnia. PE protocol (psychoeducation) begins on week 4 of treatment and both treatments overlap till week 6 when CBT-I ends and the active treatment of PE begins (i.e., imaginal and in-vivo exposures). However, CBT-I sleep diary review and sleep time adjustment will continue till the end of treatment to increase adherence
  Arms: CBTI-PE
Behavioral: Hygiene-PE — The investigators have included a non-active sleep control arm (3 Sessions)to allow for the dose response of 14 90 minute sessions. The non-active sleep control condition used in this study is a manualized protocol developed to exclude the active components of standard CBT-I treatment. Hygiene includes presentation of sleep hygiene education and reviewing daily stressors that may impact sleep before starting PE on week 4.
  Arms: Hygiene-PE

SUMMARY:
This study aims to examine whether integrating insomnia and PTSD treatment will enhance sleep, PTSD, and quality of life outcomes. This is a randomized control trial comparing integrated evidence based CBT-I into PE (CBTI-PE) versus to a non-active sleep component plus PE (hygiene-PE) to optimize PTSD, sleep, and quality of life outcomes in 90 Veterans. Such benefits would further the VA's commitment to improving the mental health, recovery, and community reintegration of Veterans detailed in the 2014-2020 VHA Strategic Plan. Findings from the proposed study offer a unique opportunity to determine the malleability of mechanisms (e.g., Total sleep time, Sleep efficiency) that can improve recovery outcomes among this vulnerable population and to inform future treatment development and research. Improved PTSD, insomnia, and quality of life outcomes can decrease risk of chronic impairment and ultimately help affected Veterans live richer, more productive lives.

DETAILED DESCRIPTION:
The lifetime prevalence of posttraumatic stress disorder (PTSD) is approximately 30% among Vietnam Veterans and 11-17% among Iraq and Afghanistan Veterans. PTSD is associated with enormous health care costs, increased suicidality, depression, poorer quality of life and functioning, physical health, and increased substance use. Prolonged exposure (PE) is an efficacious treatment for Veterans with PTSD that decreases avoidance of feared, but safe, cues. Despite PE being one of the best available treatments for PTSD, 25 to 45% of PTSD patients still meet diagnostic criteria following treatment. High rates of comorbid disorders, such as insomnia, may interfere with the efficacy of PE and limit long-term rehabilitation outcomes.

Among Veterans with PTSD, sleep disturbances are nearly universal with 70 - 87% reporting comorbid insomnia. Untreated insomnia can persist for years, is independently associated with impaired health-related quality of life, does not resolve following PTSD treatment, and can exacerbate daytime PTSD symptoms.

Importantly, insomnia may interfere with the mechanisms of PE through safety learning, habituation to feared stimuli, emotional coping, emotional processing, and cognitive abilities necessary for successful treatment.

Despite this, insomnia is not a primary intervention for Veterans with PTSD. Given these factors, it is critical to evaluate whether treating insomnia prior to PTSD will improve PTSD symptoms and quality of life outcomes. Cognitive behavioral treatment for insomnia (CBT-I) is the first line treatment of chronic and severe insomnia, which produces lasting improvements in sleep. By using CBT-I prior to, and integrated with, PE offers several novel advantages that will: 1) increase client-centered treatment by addressing the number one subjective complaint among Veterans with PTSD; 2) enhance PTSD outcomes and non-response rates by addressing insomnia-related factors that interfere with PTSD treatment; 3) act as a stepping stone and help to engage patients who are not initially willing to engage in trauma-focused PE; 4) increase rehabilitation outcomes by addressing the two leading disorders that independently affect quality of life for Veterans; 5) allow patients to address both symptoms of insomnia and PTSD within a shortened timeframe; 6) increase continuity by allowing patients to work with a single provider; and 7) decrease the risk of attrition between referral clinics and waitlists. To date, no studies have capitalized on available evidence-based CBT-I prior to PE to improve insomnia, PTSD, and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 19 years old
* Diagnosis of PTSD
* Meet diagnostic criteria for insomnia
* Enrolled at the VA San Diego Healthcare System (VASDHS) and living within 50 miles of the respective facility
* English literacy

Exclusion Criteria:

* Unmanaged psychosis or manic episodes in past year
* Substance/alcohol use disorder in past 6 months
* Diagnosed (previously or by the investigators' study screen) and untreated sleep disorder other than insomnia

  * Sleep disorders diagnosed, but stably treated, such as obstructive sleep apnea treated with continuous positive airway pressure (CPAP), will be allowed)
* Participation in concurrent psychotherapies targeting PTSD

  * Veteran can be reassessed after their PTSD treatment concludes
  * Veterans who are engaged in treatment for non-PTSD symptoms (e.g., 12-step programs) will be eligible
* Severe medical or psychiatric illness that would make it difficult to regularly attend psychotherapy sessions or participate fully in the study
* History of moderate to severe cognitive impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Colvonen, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colvonen PJ, Hunt C, Park J, Angkaw AC, Gehrman P, Clare K, Norman SB. Cognitive Behavioral Therapy for Insomnia With Prolonged Exposure Compared to Sleep Hygiene and Prolonged Exposure: A Randomized Controlled Trial. J Clin Psychiatry. 2025 Jun 4;86(3):24m15584. doi: 10.4088/JCP.24m15584. PMID 40488726
- [Derived] Park J, Hunt C, Abirgas K, Bomyea J, Colvonen PJ. Veterans who focus on sexual assault trauma show slower between-session habituation and symptom reduction during prolonged exposure treatment for posttraumatic stress disorder. Psychol Trauma. 2025 Jan;17(1):38-47. doi: 10.1037/tra0001536. Epub 2023 Jun 19. PMID 37338445
- [Derived] Lyons R, Barbir LA, Owens R, Colvonen PJ. STOP-BANG screener vs objective obstructive sleep apnea testing among younger veterans with PTSD and insomnia: STOP-BANG does not sufficiently detect risk. J Clin Sleep Med. 2022 Jan 1;18(1):67-73. doi: 10.5664/jcsm.9498. PMID 34216197

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 94 participants met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | CBTI-PE | Hygiene-PE
Started | 52 | 42
Completed | 43 (Has at least 2 timepoints to be included in ITT analyses.) | 35 (Has at least 2 timepoints to be included in ITT analyses.)
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBTI-PE | Hygiene-PE | Total
Number analyzed (Participants) | 52 | 42 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.3) | 41.2 (12.4) | 40.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 40 | 32 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 10 | 29
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 10 | 7 | 17
  White | 26 | 23 | 49
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 42 | 94
Clinician Administered PTSD Scale (CAPS) [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale. Range (0 - 80). Lower scores equate to lower PTSD severity.
  units on a scale | 38.6 (6.7) | 37 (9.5) | 38 (8.1)
Sleep Efficiency (SE) [Mean (Standard Deviation); unit: Percentage of time asleep time in bed] — Sleep Efficiency. Range (0 -100%). Higher sleep efficiency is better.
  Percentage of time asleep time in bed | 70.94 (14.46) | 74.87 (10.9) | 72.45 (13.28)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index. Range (0 - 28). Higher scores equate to worse insomnia symptoms.
  units on a scale | 21.26 (4.7) | 19.67 (4.63) | 20.53 (4.73)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Quality of Life Scores. All subscores, higher scores equate to better quality of life. Physical Health Range (7-35); Psychological Range (6-30); Social Relationships (3-15); Environment (8-40).
  units on a scale
    Physical Health | 9.38 (2.7) | 11.34 (2.09) | 10.26 (2.62)
    Psychological | 9.33 (3.28) | 11.19 (2.73) | 10.16 (3.16)
    Social relationships | 9.51 (4.04) | 11.19 (3.78) | 10.26 (4)
    Environment | 12.20 (3.27) | 13.64 (2.67) | 12.85 (3.09)

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms
Description: PTSD Symptoms will be assessed using the Clinician-Administered PTSD Scale DSM 5 (CAPS-5). Range (0 - 80). Lower scores equate to lower PTSD severity. Change in PTSD will be assessed longitudinally using linear mixed effects models of the CAPS-5 at each timepoint to estimate slope (change) over time.
Time Frame: Baseline, Post Treatment (14-weeks), Follow-up (26-weeks)
Population: Individuals who gave at least 2 time points are included in ITT analyses in the estimation models. Observed means at each timepoint are presented below.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 43 | 35
score on a scale
  Post-Treatment | 25.74 (12.34) | 28.18 (11.62)
  3 Month Follow-up | 28.59 (12.68) | 24.93 (12.61)

2. Primary Outcome: Change in Sleep Efficiency
Description: Change in sleep efficiency. Sleep efficiency is calculated from two variables acquired from daily sleep logs filled out by patient: a) time spend in bed and b) time spent asleep. Sleep efficiency = time spent asleep / time spent in bed. Range (0 -100%). Higher sleep efficiency is better. Change in Sleep Efficiency will be assessed longitudinally using linear mixed effects models of measure at each timepoint to estimate slope (change) over time.
Time Frame: Baseline, Post Treatment (14-weeks), Follow-up (26-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of time asleep time in bed
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 25 | 21
Percentage of time asleep time in bed
  Post-Treatment | 88.71 (6.46) | 78.44 (9.71)
  3 Month Follow-Up | 86.46 (7.67) | 78.23 (10.86)

3. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of life will be assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire. All subscores, higher scores equate to better quality of life. Physical Health Range (7-35); Psychological Range (6-30); Social Relationships (3-15); Environment (8-40).
Time Frame: Baseline, Post Treatment (14-weeks), Follow-up (26-weeks)
Population: Participants analyzed are the observed means. Different from the Intent to treat number of participants reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 39 | 30
score on a scale
  Physical Health - Post TX | 11.6 (5.32) | 10.53 (6.44)
  Physical Health - 3m | 10.12 (6.14) | 12.11 (7.56)
  Psychological - post treatment | 10.46 (4.81) | 10.26 (6.13)
  Psychological - 3m | 9.31 (5.77) | 11.64 (4.99)
  Social relationships - post-TX | 10.63 (5.05) | 9.49 (5.98)
  Social relationships - 3m | 9.61 (6.46) | 11.24 (4.99)
  Environment - post-tx | 12.13 (5.22) | 11.08 (6.34)
  Environment - 3m | 11.15 (6.56) | 12.94 (5.31)

4. Secondary Outcome: Change in Insomnia Severity
Description: Insomnia Severity will be assessed using the Insomnia Severity Index (ISI). Range (0 - 28). Lower scores equate to lower insomnia severity. Change in ISI will be assessed longitudinally using linear mixed effects models of the ISI scores at each timepoint to estimate slope (change) over time.
Time Frame: Baseline, week 5, Post Treatment (14-weeks), Follow-up (26-weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 45 | 36
score on a scale
  Week 5 | 15.13 (6.50) | 17.69 (4.76)
  Post-Treatment | 9.46 (6.98) | 12.93 (6.58)
  3 Month Follow-up | 11.76 (6.70) | 12.37 (7.57)

5. Other Pre Specified Outcome: The Client Satisfaction Questionnaire (CSQ)
Description: CSQ assesses client satisfaction for therapy session. Range (8-32) with higher scores equating to higher satisfaction.
Time Frame: Post Treatment ( up to 14-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 41 | 33
score on a scale | 29.41 (3.11) | 29.56 (2.97)

6. Other Pre Specified Outcome: Brief Pain Inventory
Description: Brief Pain Inventory ranges from 0 - 40, with higher score indicating worse pain.
Time Frame: post treatment, and 3-month follow-ups presented.
Population: N is for observed means only, not Intent to Treatment repeated measures analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI-PE | Hygiene-PE
Number analyzed (Participants) | 29 | 26
score on a scale
  Post-Treatment | 18.69 (9.14) | 15.63 (10.12)
  3 Month Follow-up | 18.41 (7.81) | 16.08 (9.94)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for the duration of our study ( from baseline until3-month follow-up assessment date, up to 26 weeks).
Arm/Group | CBTI-PE | Hygiene-PE
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/35
Other Adverse Events (participants affected / at risk) | 0/43 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBTI-PE (N=43) | Hygiene-PE (N=35)
Suicidal ideation (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
First, our study is limited in generalizability by an all-Veteran sample and may not fully overlap for civilians. Second, we used self-report measures of sleep. Future studies would do well to use polysomnography to capture the mechanistic effects of CBTI-PE on sleep architecture. Third, despite foundational power analyses from baseline, we were likely underpowered to capture effects of CBT-I on an active and effective treatment like PE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02774642/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02774642/SAP_001.pdf